CLINICAL TRIAL: NCT05425069
Title: Evaluation of the EEG Connectivity Using Predominantly Dexmedetomidine Anesthesia Versus Traditional TCI Propofol in Fragile Brains
Brief Title: Evaluation of the EEG Connectivity Using Predominant Dexmedetomidine as Anesthetic in Fragile Brains
Acronym: BaseDexmed
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Klinikum rechts der Isar Technische Universität München (Unknown)
Responsible Party: Principal Investigator, Pablo O. Sepulveda, DrMed Asociated Professor, Universidad del Desarrollo
Other Study IDs: Universidad Austral
Record Dates: First submitted 2022-04-16; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Aging Problems
Keywords: Frailty brain; Dexmedetomidine; Propofol; MoCA test; Frontal EEG

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dexmedetomidine with minimal concentration of propofol (D-P): Intravenous infusion with Dexmedetomidine for 10 minutes at 0.8 ug/kg/hr and so on, then induction with Propofol TCI Target 2.0 ug/ml (Schnider model) and Remifentanil TCI 4.5 ng/ml. 3 minutes after LOC Propofol will be reduced to 0.5 ug/ml. intubate using Remifentanil 4.5 ng/ml and Rocuronio 0.5 mg/kg.
  Anesthesia will be dynamically adjusted to maintain SEF95 remains at minimum values at 10 Hz for the rest of the surgery. Sedline will be maintained for up to 60 min post-op. in the recovery room. Data will be retrieved via pen drive stick from SEdline
  Interventions: Drug: Comparison MoCA test and EEG connectivity pre, intra and postoperative between groups P vs D-P
- Propofol TCI fine titrated (P): Basal frontal EEG with eyes opened and closed (90 sec each) The previous bolus of Lidocaine in a 20 mg intravenous dose, TCI Propofol Induction (Schnider Model) is initiated starting 8 mg/kg/h until clinical unconsciousness (LOC loss of response to the call and to moderate stimulus in the shoulder) and then it is passed to TCI to keep the Ce calculated to the LOC.
  After LOC, we proceed to intubate using Remifentanil 4.5 ng/ml and Rocuronio. Anesthesia will be dynamically adjusted to maintain Sedline SEF 95 value of minimum at 10Hz. Sedline will be maintained for up to 60 min post LOC in the recovery room.
  Data will be retrieved via pen drive stick.
  Interventions: Drug: Comparison MoCA test and EEG connectivity pre, intra and postoperative between groups P vs D-P

INTERVENTIONS:
Drug: Comparison MoCA test and EEG connectivity pre, intra and postoperative between groups P vs D-P — We compare de impact in EEG, anesthetic condition, and recovery EEG and cognitive clinical characteristic with MoCA test between both groups (propofol vs propofol dexmedetomidine)
  Other Names: comparison EEG evolution between study groups

SUMMARY:
Elderly brains that present a lower intrinsic cortical activity are very dependent on arousal feeding. In these patients, a strong blockade of afferences generates a synchronic state with a high tendency to sleep. This is done with drugs such as Dexmedetomidine and its indirect effect of inhibiting the amplification of signals and opioids such as remifentanil. Then, by adding a micro-dose of a gabaergic substance to induce loss of consciousness, unconsciousness would be maintained due to the low requirement of a fragile and synchronous brain by a slow continuous injection of an alpha2 agonist. In previous experience, doses of about one-fifth of the usual would be sufficient to maintain unconsciousness (or perhaps disconnected consciousness that could be useful in avoiding excessive depression in slowed integration pathways). These patients also present deficits in the orexinergic response that manifest themselves in greater neuronal inertia and delayed awakening. Gabaergic drugs (propofol and sevoflurane) are especially depressing to orexinergic nuclei.

This approach to the elderly brain could have an impact on recovering more easily connectivity of those CNC networks.

In elderly patients, one aspect that could control the phenomena of altered connectivity and its impact in developing delirium is the limitation of connection with the environment before the capacity of integration of cortical information has been completely recovered. To analyze frontoparietal connectivity, front frontal coherence, phase lag index, or similar it is necessary to a multichannel EEG (e.g. 10 channels). Otherwise, the frontal EEG from the SEDline monitor device allowed to analyze only spectral characteristics (power, peak frequency, etc.) and correlate them with clinical observations (MoCA).

DETAILED DESCRIPTION:
Research question: Does subcortical drug-based anesthesia allow better recovery of consciousness (integration of information) than the classic gabaergic drug-based technique in elderly and fragile brains?

Primary hypothesis: The anesthetic technique based on subcortical anesthesia with Dexmedetomidine and Remifentanil and minimal gabaergic doses (Propofol) allow fragile and slower brains a faster recovery of cortical connectivity. This behavior represents part of the evidence of neural inertia in sleep and anesthesia.

Objectives:

1. Primary: Evaluation of the normalization of the frontal EEG of patients with mostly subcortical anesthesia (Dexmedetomidine-Remifentanil.-low Propofol in TCI ) or classic technique (Remifentanil-Propofol in TCI) versus its preoperative basal control.
2. Secondary:

   1. To estimate the recovery of the cognitive condition with MoCA test, agitation scale, and delirium CAM-ICU.
   2. To identify behavioral patterns of the EEG with two different anesthetic techniques

Participants

1. Target population: Patients scheduled for elective surgery, any sex, non-neurological procedure lasting more than 60 minutes, who do not meet the exclusion criteria.
2. Eligibility criteria Inclusion criteria: - ASA I - II - Age: over 70 years old

Exclusion criteria:

* Neurological, or systemic disease that affects the central nervous system in a secondary way
* Abnormal admission neurological physical exam
* Consumption of benzodiazepines, tricyclic antidepressants, sympathomimetics, modafinil, opioid analgesics, histaminergic, antihistamines, cholinergic, anticholinergics, dopaminergic, antidopaminergic, and antihypertensive with alpha-agonist effect in the last 48 hours.
* History of adverse or allergic reactions to Propofol (allergy to soy or any other component of it)
* History of alcohol or drug abuse
* Subjects with "fast sequence induction" indication

Withdrawal criteria:

* Patients presenting with any adverse event during induction (excitation, hypotension, bradycardia <40 x min, nausea).
* Subsequent refusal to participate in the study

  1. Randomize patients into two groups of a similar number of individuals. Group 1: Propofol TCI - Remifentanil anesthesia. TCI Propofol (Schnider PKPD model), 5-minute step-by-step induction. After LOC stay in this calculated effect site concentration, add Remifentanil TCI PKPD model Minto target 4.5 ng/ml, Rocuronium intubation dose. EEG Sedline monitoring all the surgery until 1 hour postoperatively Group 2: Dexmedetomidine 0.8 ug/kg/h during 10 minutes- then Propofol TCI target 2 ug/ml (Schnidel model) during 3 min and reduce to 0.5 ug/ml, Remifentanil TCI (PK model Minto), after LOC Rocuronium intubation dose. EEG Sedline monitoring all the surgery until 1 hour postoperatively 0,5 ug/ml after LOC
  2. Both groups were evaluated with MoCA and CAMICU tests: Pre-operative and post-operative cognitive assessments will be performed with MoCA test and CAMICU test, which will be correlated with the EEG characteristics of each group both in the baseline measurements, intraoperative behavior, and after one hour in the recovery room
  3. Basal frontal EEG with eyes opened and closed (90 sec each) preoperatively without any drug effect

To protect the risk of awareness or excess of EEG depression, during surgery, Anesthesia will be dynamically adjusted to maintain SEF95 remains at minimum values at 8-10 Hz for the rest of the surgery.

Sedline will be maintained for up to 60 min post-op. in the recovery room. Data will be retrieved via pen drive stick (edf data corresponding to raw EEG) and other trends data of the Sedlie monitor using the proprietary software Masimo Instrument Configuration Tools

In both groups, the Systolic Blood Pressure, Freq. Cardiac, Pulse Oximetry, Capnography, and Sedline EEG will be monitored throughout the surgical procedure and for at least one hour postoperatively. No drugs such as ketamine, midazolam, atropine, or other anticholinergics will be used at any time.

Hemodynamics will be supported with volume, ephedrine, or phenylephrine according to the criteria of the anesthesiologist.

Unexpected events during the induction: Any anesthetic induction has risks of hemodynamic instability, arrhythmias, and respiratory apneas. Most of them are easy to handle anesthesiological based on volume, vasoactive drugs such as ephedrine, and respiratory assistance.

In this case, a minimum or no incidence of these is expected because healthy patients are included.

Exceptional situations such as anaphylactic reactions to propofol (very rarely described) will be cause for suspension of the case study and treated with usual protocols for the case.

During the Surgery, the analgesic requirement will be adjusted with Remifentanil TCI concentration in the clinical criterium of the anesthetist.

Postoperative analgesia will be multimodal, with or without regional block depending on the anesthetist's criterium and type of surgery.

Database and data management: SEDLINE data is retrieved online by proprietary software to a PC. These, together with the manual control data, will be collected in a Microsoft Excel 2011 worksheet and exported to a STATA 10 statistical program template, with which the analysis will be performed.

A work together with the Basic Data Manager of the Anesthesia Service to safeguard the information and its confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria Inclusion criteria
* surgery over 60 min
* ASA I - II
* Age: over 70 years old

Exclusion Criteria:

* - Neurological, or systemic disease that affects the central nervous system in a secondary way
* Abnormal admission neurological physical exam
* Consumption of benzodiazepines, tricyclic antidepressants, sympathomimetics, modafinil, opioid analgesics, histaminergic, antihistamines, cholinergic, anticholinergics, dopaminergic, antidopaminergic, and antihypertensive with alpha-agonist effect in the last 48 hours.
* History of adverse or allergic reactions to Propofol (allergy to soy or any other component of it)
* History of alcohol or drug abuse
* Subjects with "fast sequence induction" indication

Withdrawal criteria:

* Patients presenting with any adverse event during induction (excitation, hypotension, bradycardia <40 x min, nausea).
* Subsequent refusal to participate in the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients over 70 years, programmed to elective surgery longer than 60 min
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of both groups in Recovery Cognitive and electroencephalogram EEG Conditions, during and after surgery | pre, intra and one hour postoperative in recovery room
  Measuring instruments: Cognitive MoCA test (Montreal Cognitive assessment) pre and one-hour post-operative.
  Drug consumption to maintain a Spectral Edge Frequency SEF 95 over 10Hz as calculated Propofol effect-site concentration using Schnider PKPD model.
  Evaluation of basal alpha power preop, at the loss of response time, during de surgery every 20 minutes, and during the first-hour post operatively (in dB)
  * Neurological milestones: Montreal Cognitive assessment MoCA test pre and one-hour post-op
  * Anesthetic depth: SEDLINE® spectrogram dynamic during anesthetic all process and one hour after using the Patient state Index, the Spectral edge frequency 95, the alpha band power, the existence of Burst suppression,
  * Basic monitoring: Electrocardiogram ECG, non-invasive BP, pulse oximetry, and capnography.
Presence of post operative delirium and agitation | post operative in recovery room, and late one week
  evaluated by sedation-agitation scale SAS every 30 min, and confusion assessment method CAM ICU scale every 30 min

SECONDARY OUTCOMES:
Postopertive pain | in Recovery room evolution
  Using the Visual Analog Scale VAS

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Sepulveda V., Dr. Med, Principal Investigator — iversidad Austral, Sevicio de salud Valdivia
Locations (1):
- Hospital Base San Jose, Osorno, Los Lagos Region, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Publishing in a peer-review journal